CLINICAL TRIAL: NCT02236299
Title: Diastolic RV EvAluation With Millar Catheter to Investigate the Effect of Glucagon-Like Peptide-1 (GLP-1) on Right Ventricular Function During Elective Coronary Angioplasty and Stenting - DREAM GLP-1
Brief Title: Diastolic RV EvAluation With Millar Catheter to Investigate the Effect of Glucagon-Like Peptide-1 (GLP-1) on Right Ventricular Function During Elective Coronary Angioplasty and Stenting
Acronym: DREAM GLP-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01851
Record Dates: First submitted 2014-06-23; First posted 2014-09-10 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Right Coronary Artery Percutaneous Coronary Intervention; Right Ventricular Diastolic Dysfunction
Keywords: Right Coronary Artery; Percutaneous Coronary Intervention; Diastolic Dysfunction; Glucagon-like peptide-1; GLP-1; Stunning; Cardioprotection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- saline placebo infusion (Placebo Comparator): 30 minute infusion of a saline placebo Right coronary artery percutaneous coronary intervention
  Interventions: Procedure: Right Coronary Artery Percutaneous Coronary Intervention; Other: saline placebo infusion
- GLP-1 infusion (Experimental): 30 minute infusion of GLP-1 Right coronary artery percutaneous coronary intervention
  Interventions: Procedure: Right Coronary Artery Percutaneous Coronary Intervention; Other: GLP-1 Infusion

INTERVENTIONS:
Procedure: Right Coronary Artery Percutaneous Coronary Intervention
  Other Names: Device - stent
Other: saline placebo infusion — 30 minute placebo infusion used as a comparator to the GLP-1 infusion
  Arms: saline placebo infusion
Other: GLP-1 Infusion — 30 minute infusion GLP-1
  Arms: GLP-1 infusion

SUMMARY:
The heart requires nutrients and oxygen carried in the blood to generate energy for healthy pump function. Blood is supplied via heart vessels called coronary arteries. When the arteries narrow the investigators call this coronary artery disease. Narrowing and blockage of the coronary arteries can cause chest pain (angina), breathlessness (due to a reduction in pump function) and if prolonged even irreversible muscle damage known as a heart attack. The investigators can treat patients with coronary artery disease with drugs that reduce the workload on the heart or with balloons and hollow metal tubes (stents) to open the narrowed coronary arteries and improve the blood supply. These treatments can relieve angina, improve breathlessness and avert heart muscle damage during a heart attack. A potential new mechanistic effect is emerging by modulating the type of fuel used by the heart to generate energy more efficiently has been tested in the left ventricle. This study is designed to see if mechanistic effect provides the same protection in the right ventricle. It is hoped that this may further improve heart pump function and reduce the size of a heart attack in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Able to give informed consent
* Elective percutaneous intervention for a single vessel right coronary artery stenosis >75%
* Normal right ventricular function

Exclusion Criteria:

* Severe co-morbidity expected life (<6months)
* Nicorandil or a GLP-1 receptor agonist or DPP-4 inhibitor use
* Women of child bearing age
* Myocardial infarction within the previous 3 months
* Previous coronary artery bypass graft to the RCA
* Significant known left to right shunt
* Permanent pacemaker
* Atrial fibrillation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Improvement in RV diastolic dysfunction (Tau, dP/dt min) between control and GLP-1 groups. | Change betweeen Balloon Occlusion One (Baseline) and Balloon Occlusion Two (30 minutes later)
  Tau - the time constant of diastolic relaxation is a sensitive measure of ventricular function.
  Control Group - 15 patients are randomised to receive a placebo saline infusion.
  GLP-1 Group - 15 patients are randomised to receive a GLP-1 infusion.
  Balloon Occlusion One - is performed at the start of the procedure and is a measure of baseline ventricular function.
  Balloon Occlusion Two - is performed directly after a 30 minute infusion of either the saline control or GLP-1.
  All measurements are performed while the patient is in the catheter laboratory.

SECONDARY OUTCOMES:
Improvement in RV systolic function (EF, dP/dt max), between control and GLP-1 groups. | Change betweeen Balloon Occlusion One (Baseline) and Balloon Occlusion Two (30 minutes later)
  EF - the Ejection Fraction is the percentage of blood ejected by the ventricle and is considered as a sensitive measure of ventricular function.
  Control Group - 15 patients are randomised to receive a placebo saline infusion.
  GLP-1 Group - 15 patients are randomised to receive a GLP-1 infusion.
  Balloon Occlusion One - is performed at the start of the procedure and is a measure of baseline ventricular function.
  Balloon Occlusion Two - is performed directly after a 30 minute infusion of either the saline control or GLP-1.
  All measurements are performed while the patient is in the catheter laboratory.
Collaterals and microcirculatory differences between control and GLP-1 groups | Change betweeen Balloon Occlusion One (Baseline) and Balloon Occlusion Two (30 minutes later)
  Control Group - 15 patients are randomised to receive a placebo saline infusion.
  GLP-1 Group - 15 patients are randomised to receive a GLP-1 infusion.
  Balloon Occlusion One - is performed at the start of the procedure and is a measure of baseline ventricular function.
  Balloon Occlusion Two - is performed directly after a 30 minute infusion of either the saline control or GLP-1.
  All measurements are performed while the patient is in the catheter laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Hoole, BM BCh, MA, MD, Study Chair — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital NHS Foundation Turst, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Background] Read PA, Hoole SP, White PA, Khan FZ, O'Sullivan M, West NE, Dutka DP. A pilot study to assess whether glucagon-like peptide-1 protects the heart from ischemic dysfunction and attenuates stunning after coronary balloon occlusion in humans. Circ Cardiovasc Interv. 2011 Jun;4(3):266-72. doi: 10.1161/CIRCINTERVENTIONS.110.960476. Epub 2011 May 17. PMID 21586690